CLINICAL TRIAL: NCT05173376
Title: Socioeconomic Position and the Effect of Portion Size Reduction: a 1-day Dietary Behaviour Experimental Study
Brief Title: SEP and the Impact of Portion Size on Daily Energy Intake
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Liverpool (Other)
Collaborators: European Research Council (Other)
Responsible Party: Principal Investigator, Eric Robinson, Principal Investigator (Reader in Psychological Sciences), University of Liverpool
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: 803194
Record Dates: First submitted 2021-10-14; First posted 2021-12-29 (Actual); Last update posted 2023-01-10 (Actual); Status verified 2023-01

CONDITIONS: Diet, Healthy; Eating Behavior; Obesity
Keywords: portion size; socio-economic position; eating behaviour
MeSH Terms: conditions — Feeding Behavior; Obesity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Larger portions (Experimental): the main meal component (lunch/dinner) served to participants in the laboratory, reflecting 100% portion. All other foods are identical across conditions (e.g. sides, seconds, breakfast, dessert, snacks).
  Interventions: Behavioral: Portion size manipulation
- Smaller portions (Experimental): the main meal component (lunch/dinner) served to participants in the laboratory, reflecting 66% portion (i.e. reduced portion size). All other foods are identical across conditions (e.g. sides, seconds, breakfast, dessert, snacks).
  Interventions: Behavioral: Portion size manipulation

INTERVENTIONS:
Behavioral: Portion size manipulation — The intervention was administered via changing portion sizes of foods served to participants.

SUMMARY:
Reducing food portion size is a potential strategy to reduce energy intake. There is some evidence to suggest that individuals with lower socioeconomic position (SEP) intend to eat more from larger portions, suggesting that the effect of portion size on food intake might vary by SEP. However, no study has tested this by measuring actual food intake. This study examines whether reductions to the portion size of components of a main meal will reduce daily energy intake, and whether and how socioeconomic position (higher vs lower) moderates the portion size effect.

In a crossover experiment, participants will be served all meals in the lab on two separate days, with the portion size of main meal components at lunch and dinner manipulated (i.e. smaller on one day vs larger on the other day). All other foods offered are identical. Food intake from the portion-manipulated lunch and dinner, as well as all other meal components (breakfast, dessert, seconds, snacks) will be measured, and any additional food consumed by the participant will be measured using self-report, giving total daily energy intake (kcal).

DETAILED DESCRIPTION:
See attached protocol document.

ELIGIBILITY:
Inclusion Criteria:

* Female
* UK (United Kingdom) residents, aged 18 or over
* Fluent in English
* willing to consume the test foods
* Self report liking of test foods
* BMI between 22.5 - 32.5kg2

Exclusion Criteria:

* taking medication which affects appetite
* currently pregnant
* history of eating disorders
* currently on a diet to lose weight
* food allergies, intolerances or specific dietary requirements (including being vegetarian or vegan)
* participated in 2018 Mood Study
* currently participating in another study where meals are provided

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Identify as female
Enrollment: 54 (Actual)
Dates: Start 2021-10-25 (Actual); Primary Completion 2022-04-07 (Actual); Study Completion 2022-04-07 (Actual)

PRIMARY OUTCOMES:
Daily energy intake | 24 hours after intervention administered
  Total energy (kcal) consumed from breakfast, lunch, dinner, dessert, snackbox, and any self-reported additional foods.

SECONDARY OUTCOMES:
Appetite | 24 hours after intervention administered
  Hunger and fullness sensations before and after laboratory-based meals (self-reported on visual analogue scales anchored at 0 'Not at all' and 100 'Extremely')
Moderate-vigorous physical activity | 24 hours after intervention administered
  Moderate-vigorous physical activity (recorded using wearable activity tracker), operationalised as active minutes/day (logged for activities with a metabolic equivalent of >/3)

CONTACTS AND LOCATIONS:
Overall Officials: Eric Robinson, PhD, Principal Investigator — Study Principle Investigator
Locations (1):
- University of Liverpool, Liverpool, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Study data (anonymised) will be shared on the Open Science Framework (OSF)
Supporting Information: Study Protocol, SAP
Time Frame: On publication, indefinitely
Access Criteria: Open website
URL: https://osf.io/scjn6/

REFERENCES:
- [Derived] Langfield T, Clarke K, Marty L, Jones A, Robinson E. Socioeconomic position and the influence of food portion size on daily energy intake in adult females: two randomized controlled trials. Int J Behav Nutr Phys Act. 2023 Apr 27;20(1):53. doi: 10.1186/s12966-023-01453-x. PMID 37101143
- Available data/document: Study Protocol — https://osf.io/scjn6/ — Protocol on the Open Science Framework (OSF)
- Available data/document: Statistical Analysis Plan — https://osf.io/scjn6/
- Available data/document: Individual Participant Data Set — https://osf.io/scjn6/ — The study protocol and statistical analysis plan were pre-registered on the OSF prior to starting recruitment. Participant dataset (anonymised) will be made available when results are published.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-10-01): https://cdn.clinicaltrials.gov/large-docs/76/NCT05173376/Prot_SAP_000.pdf